CLINICAL TRIAL: NCT03452098
Title: Examination and Post-operative Rehabilitation of University Athletes With Osteochondral Lesions of the Knee: A Case Series Report
Brief Title: Post-Operative Rehabilitation of Knee Osteochondral Defect: A Case Series
Status: Completed | Type: Observational
Sponsor: California State University, Northridge (Other)
Responsible Party: Sponsor
Other Study IDs: IRB-FY18-11
Record Dates: First submitted 2018-02-09; First posted 2018-03-02 (Actual); Last update posted 2019-02-11 (Actual); Status verified 2019-02

CONDITIONS: Osteochondral Defect; Osteochondritis Dissecans
MeSH Terms: conditions — Osteochondritis Dissecans

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A case-series review was performed on five collegiate athletes with osteochondral lesions of the knee at California State University, Northridge (CSUN). All subjects received surgical intervention to treat the defect. The surgeries performed were either an Osteoarticular Transfer System (OATS) procedure and/or a Microfracturing procedure. Subjects were treated post-operatively by the CSUN team physical therapist and/or athletic trainers at CSUN. This paper seeks to provide information about osteochondral defects of the knee, the surgical interventions, and a protocol for post-operative treatment and rehabilitation of such injuries.

ELIGIBILITY:
Inclusion Criteria:

* Student athlete at CSUN
* Diagnosed with Osteochondral dissecans (OCD)
* Underwent surgical procedure to treat OCD
* Treated postoperatively by the team physical therapist and/or athletic trainers at CSUN.

Exclusion Criteria:

- No concurrent ligamentous injures to the knee during the time of subject participation in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The subjects were recruited from a population of student athletes at California State University, Northridge. These athletes were being treated by the Physical Therapy and/or Athletic Training Departments for Osteochondral Defect of the knee.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Level of Function | Through study completion; an average of 6 months
  Determined by subject's ability to return to play of his/her respective sport

SECONDARY OUTCOMES:
Pain | Monthly until the completion of the study; an average of 6 months
  Pain as measured by the Visual Analog Scale (VAS), 0 (No pain) - 10 (Severe Pain)

CONTACTS AND LOCATIONS:
Overall Officials: Aimie Kachingwe, PT, DPT, EdD, OCS, FAAOMPT, Principal Investigator — CSUN Physical Therapy Department
Locations (1):
- California State University, Northridge, Northridge, California, United States